CLINICAL TRIAL: NCT02571595
Title: Efficacy Potential of an Internet-based Sleep Program to Improve Sleep Quality in People With HIV
Brief Title: A Sleep Program to Improve Sleep Quality in People With HIV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Sleepio (Industry)
Responsible Party: Principal Investigator, Lesley K. Fellows, Neurologist, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14-368-BMB; CTN S 290 (Other: CIHR Canadian HIV Trials Networ)
Record Dates: First submitted 2015-08-25; First posted 2015-10-08 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: HIV - Human Immunodeficiency Virus; Insomnia Disorder
Keywords: HIV - Human Immunodeficiency Virus; digital cognitive behavioural therapy for insomnia (dCBT-I); insomnia; cognitive Impairment; concentration; productivity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate dCBT-I group (Experimental): Digital cognitive behavioural therapy for insomnia (dCBT-I) is a 6 session training program (spanning 6 to 12 weeks) designed to improve sleep. Participants in the immediate dCBT-I group will receive the Sleepio intervention shortly after enrollment.
  Interventions: Behavioral: Digital cognitive behavioural therapy for insomnia (dCBT-I)
- Waitlist control group (Experimental): Participants in the waitlist control group will receive sleep hygiene recommendations from validated online resources for HIV patients (http://www.catie.ca/en/positiveside/winter-2013/sleep-tight) around the time of enrollment. They will start the digital cognitive behavioural therapy for insomnia (dCBT-I) intervention 12-14 weeks after the initial enrollment.
  Interventions: Behavioral: Digital cognitive behavioural therapy for insomnia (dCBT-I)

INTERVENTIONS:
Behavioral: Digital cognitive behavioural therapy for insomnia (dCBT-I) — dCBT-I is a computer-based treatment intervention that provides strategies to improve sleep and daytime function (concentration, productivity) in individuals with insomnia
  Other Names: Sleepio

SUMMARY:
Sleep problems, such as insomnia, are more frequent and intense in individuals living with HIV. These sleep difficulties can increase the difficulties in thinking and concentrating. Digital cognitive behavioral therapy for insomnia (dCBT-I) is a computer-based treatment intervention that provides strategies to improve sleep. This intervention has been shown to improve sleep and daytime function (concentration, productivity) in people with insomnia. However, the effects of this intervention in people living with HIV are unknown.

DETAILED DESCRIPTION:
Sleep disturbances have been consistently reported in HIV+ individuals, and occur early in the course of infection. Among disorders of sleep commonly found in HIV, insomnia is by far the most frequent condition, affecting almost 75% of HIV-infected individuals. Compared to non-infected individuals, HIV+ patients are 17% more likely to develop insomnia. Furthermore, not only is insomnia more frequent in HIV; it is also more severe in HIV+ compared to HIV- individuals. The precise mechanisms underlying the vulnerability of this population to insomnia still remain hypothetical, and might involve neurodegenerative processes related to the infection, associated mood disorders (e.g., depression, anxiety), side effects of antiretroviral medications, and psychosocial factors. Importantly, sleep disorders in HIV have been demonstrated to affect the severity of the infection. For instance, sleep disturbances were shown to mediate the association between psychological distress and immune status (T-cytotoxic/suppressor cell counts). In addition, sleep disruption also affects responses to treatment, as illustrated by a report demonstrating that sleep disturbances mediate the association between medication adherence and self-reported HIV symptom severity. Finally, insomnia in HIV seems to be closely associated with the presence of cognitive disturbances. Indeed, virtually all HIV infected individuals with cognitive impairment present insomnia complaints, and greater sleep disturbances were associated with worse cognitive performance (e.g., executive functions, psychomotor speed) in this population. Therefore, insomnia has been shown to affect symptom severity, treatment adherence and cognition in HIV+ individuals.

Despite this demonstrated importance of sleep for the well-being of HIV patients, there are very few studies of sleep treatment interventions in HIV. Two studies have implemented an educational intervention promoting healthy sleep habits (e.g., healthy diet, reduced caffeine consumption, no exercise before bedtime, regular sleep-wake schedules), consisting of either one single session or 10 weekly sessions, with little or no consistent sleep improvement in this population. This is not surprising given that previous studies showed the very limited efficacy of interventions focusing solely on sleep hygiene in a general chronic insomnia population.

The most effective treatment for chronic insomnia currently consists of a multimodal psychological intervention, called cognitive-behavioral therapy for insomnia (CBT-I). CBT-I improves sleep to the same degree as hypnotic medications in the short term, but, in contrast to hypnotics, shows no side effects and remains effective in the long term, with sustained improvement in sleep and daytime functioning up to 2 years after completion of the therapy. CBT-I has proven effective in patients with primary insomnia (i.e. without associated medical condition), as well as in insomnia comorbid with depression or cancer. However, the efficacy of CBT-I has not been studied in HIV+ individuals with insomnia.

Digital Cognitive-Behavioural Therapy for Insomnia (CBT-I): the Sleepio program

CBT-I is an intervention aimed at breaking the patterns of maladaptive thinking and behavior that serve to maintain insomnia. It includes a range of techniques including a behavioral component (stimulus control, sleep restriction, relaxation) combined with a cognitive (managing sleep related worries, the racing mind and intrusive thoughts) and an educational (sleep hygiene) component. CBT-I is usually dispensed in group sessions, including 5 to 8 patients and a trained therapist. The different components of CBT-I are then covered in 6 to 8 weekly sessions of 60-90 minutes each. While CBT-I has been demonstrated as an efficacious treatment option, the personnel-intensive nature of CBT-I constitutes an important barrier to widespread clinical use.

Web-based (digital) CBT-I has been developed to overcome this barrier. Two randomized controlled trials (RCT) have evaluated separate digital CBT-I (dCBT-I) applications. In a first study, a six-week wait-list controlled trial of self-help dCBT-I was tested via a simple web-based platform delivering CBT-I content. Insomnia improvement was significantly better in the dCBT-I group when compared to wait-list control, at 4 weeks follow-up. In addition, 48 weeks following the intervention, within-subjects improvements in insomnia severity were also observed. The second RCT of CBT-I included a six-week placebo-controlled dCBT-I intervention, using a media rich, interactive application with an online discussion forum for users. This platform, named Sleepio (www.sleepio.com), allowed users to receive weekly, interactive sessions with an online virtual therapist. That RCT showed large effects on sleep efficiency (d=1.00) and insomnia severity (using the Sleep Condition Indicator (SCI) scale, d= .77), relative to the placebo control, at 8 week follow-up. Overall more than 75% of patients responded to the intervention, as defined by the recovery of healthy sleep efficiency levels. In addition, dCBT-I also significantly improved daytime function, including self-reported assessment of concentration and productivity, thereby suggesting a potential benefit of CBT-I for cognitive functions.

The current intervention sub-study will test the Sleepio dCBT-I intervention in people with HIV. Free access will be provided to the Sleepio program. The program will be delivered entirely online, in 6 weekly sessions spread over 6-12 weeks. The CBT-I sessions will be delivered by an animated virtual therapist, "The Prof". At the start of therapy, participants will complete a short questionnaire, which will be used to suggest examples of goals. Participants will be encouraged to complete a daily sleep diary online throughout the entire course, which will be used to provide personalized help. Indeed, all interactions with the virtual therapist will be dynamically driven by information from daily sleep diaries completed by the user, to provide baseline, adherence, performance and progress data; sleep diary information will also be used to tailor sleep restriction schedules as a function of to the patients' usual bedtimes. Within each therapy session, sleep diary data will be reviewed, goals will be reviewed and new targets will be set. The treatment content will be based on CBT for insomnia manuals and includes the following techniques: psycho-education, goal setting, sleep hygiene, sleep restriction, stimulus control, cognitive restructuring, paradoxical intention, mindfulness, positive imagery, relaxation (progressive muscle relaxation & autogenic training), putting the day to rest, thought stopping. Participants will be encouraged to select an appointment time for the Sleepio session and will be prompted via email if they do not attend. In addition, participants will receive an email reminder each morning to prompt them to fill in their sleep diary and will have access to a moderated online community and an online library of information about sleep throughout the course of the intervention. They will be able to view their online 'case file' which includes four sections: a progress review, a reminder of strategies to try out in between sessions, an agreed sleep schedule and a list of further reading. In addition to the Sleepio program, participants will be asked to complete a short set of questionnaires assessing mood, quality of life, cognitive symptoms and sleep quality via an online link prior at the start and end of the program, and at their next routine (main study) follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of insomnia disorder (Sleep Condition Indicator [SCI] ≤ 16)
* Able to have convenient weekly access to the Internet
* Stable medical condition
* Have been on a stable HAART regimen for > 6 months
* Have not had a change in medications that could potentially interfere with sleep or cognition in the past 4 months.

Exclusion Criteria:

* Berlin questionnaire score indicating high risk of obstructive sleep apnea
* Known history of sleep disorders (e.g., narcolepsy, hypersomnia, restless legs syndrome, REM-sleep behavior disorder) which currently require or previously required treatment
* Ongoing involvement in night shift work
* Not able to complete the 12 weeks of the sleep intervention due to a scheduling conflict

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Ratio of total sleep time over time in bed | 12 weeks
  Obtained from the online self-reported sleep diaries aggregated over 7 days, completed at study entry and again at 12 weeks

SECONDARY OUTCOMES:
Insomnia Severity as assessed by the Insomnia Severity Index | 12 weeks
  Obtained from the online self-reported questionnaire completed at study entry and again at 12 weeks
Cognitive performance as assessed by the Brief Cognitive Ability Measure (B-CAM) | 9 months
  Ruler-like measure of cognitive ability combining self-report and performance items
Anxiety and Depression symptoms as assessed by the Hospital Anxiety Depression Scale | 9 months
  Questionnaire
Quality of life as assessed by the WHO-QOL-HIV | 9 months
  Questionnaire
Quality of life as assessed by the EQ-5D | 9 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lesley K Fellows, MD, DPhil, Principal Investigator — McGill University
Locations (1):
- Montreal Neurological Institute and Hospital (McGill University), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized individual data may be requested from the investigators.

REFERENCES:
- [Background] Norman SE, Chediak AD, Kiel M, Cohn MA. Sleep disturbances in HIV-infected homosexual men. AIDS. 1990 Aug;4(8):775-81. doi: 10.1097/00002030-199008000-00009. PMID 2261133
- [Background] Rubinstein ML, Selwyn PA. High prevalence of insomnia in an outpatient population with HIV infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Nov 1;19(3):260-5. doi: 10.1097/00042560-199811010-00008. PMID 9803968
- [Background] Jean-Louis G, Weber KM, Aouizerat BE, Levine AM, Maki PM, Liu C, Anastos KM, Milam J, Althoff KN, Wilson TE. Insomnia symptoms and HIV infection among participants in the Women's Interagency HIV Study. Sleep. 2012 Jan 1;35(1):131-7. doi: 10.5665/sleep.1602. PMID 22215927
- [Background] Low Y, Goforth HW, Omonuwa T, Preud'homme X, Edinger J, Krystal A. Comparison of polysomnographic data in age-, sex- and Axis I psychiatric diagnosis matched HIV-seropositive and HIV-seronegative insomnia patients. Clin Neurophysiol. 2012 Dec;123(12):2402-5. doi: 10.1016/j.clinph.2012.05.004. Epub 2012 Jun 23. PMID 22727712
- [Background] Cruess DG, Antoni MH, Gonzalez J, Fletcher MA, Klimas N, Duran R, Ironson G, Schneiderman N. Sleep disturbance mediates the association between psychological distress and immune status among HIV-positive men and women on combination antiretroviral therapy. J Psychosom Res. 2003 Mar;54(3):185-9. doi: 10.1016/s0022-3999(02)00501-9. PMID 12614827
- [Background] Babson KA, Heinz AJ, Bonn-Miller MO. HIV medication adherence and HIV symptom severity: the roles of sleep quality and memory. AIDS Patient Care STDS. 2013 Oct;27(10):544-52. doi: 10.1089/apc.2013.0221. Epub 2013 Sep 13. PMID 24032625
- [Background] Gamaldo CE, Gamaldo A, Creighton J, Salas RE, Selnes OA, David PM, Mbeo G, Parker BS, Brown A, McArthur JC, Smith MT. Evaluating sleep and cognition in HIV. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):609-16. doi: 10.1097/QAI.0b013e31829d63ab. PMID 23722610
- [Background] Hudson AL, Portillo CJ, Lee KA. Sleep disturbances in women with HIV or AIDS: efficacy of a tailored sleep promotion intervention. Nurs Res. 2008 Sep-Oct;57(5):360-6. doi: 10.1097/01.NNR.0000313501.84604.2c. PMID 18794720
- [Background] Webel AR, Moore SM, Hanson JE, Patel SR, Schmotzer B, Salata RA. Improving sleep hygiene behavior in adults living with HIV/AIDS: a randomized control pilot study of the SystemCHANGE(TM)-HIV intervention. Appl Nurs Res. 2013 May;26(2):85-91. doi: 10.1016/j.apnr.2012.10.002. Epub 2012 Dec 21. PMID 23265919
- [Background] Morin CM. Cognitive-behavioral approaches to the treatment of insomnia. J Clin Psychiatry. 2004;65 Suppl 16:33-40. PMID 15575803
- [Background] Morin CM, Hauri PJ, Espie CA, Spielman AJ, Buysse DJ, Bootzin RR. Nonpharmacologic treatment of chronic insomnia. An American Academy of Sleep Medicine review. Sleep. 1999 Dec 15;22(8):1134-56. doi: 10.1093/sleep/22.8.1134. PMID 10617176
- [Background] Morin CM, Vallieres A, Guay B, Ivers H, Savard J, Merette C, Bastien C, Baillargeon L. Cognitive behavioral therapy, singly and combined with medication, for persistent insomnia: a randomized controlled trial. JAMA. 2009 May 20;301(19):2005-15. doi: 10.1001/jama.2009.682. PMID 19454639
- [Background] Riemann D, Perlis ML. The treatments of chronic insomnia: a review of benzodiazepine receptor agonists and psychological and behavioral therapies. Sleep Med Rev. 2009 Jun;13(3):205-14. doi: 10.1016/j.smrv.2008.06.001. Epub 2009 Feb 7. PMID 19201632
- [Background] Morin CM, Colecchi C, Stone J, Sood R, Brink D. Behavioral and pharmacological therapies for late-life insomnia: a randomized controlled trial. JAMA. 1999 Mar 17;281(11):991-9. doi: 10.1001/jama.281.11.991. PMID 10086433
- [Background] Manber R, Edinger JD, Gress JL, San Pedro-Salcedo MG, Kuo TF, Kalista T. Cognitive behavioral therapy for insomnia enhances depression outcome in patients with comorbid major depressive disorder and insomnia. Sleep. 2008 Apr;31(4):489-95. doi: 10.1093/sleep/31.4.489. PMID 18457236
- [Background] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part I: Sleep and psychological effects. J Clin Oncol. 2005 Sep 1;23(25):6083-96. doi: 10.1200/JCO.2005.09.548. PMID 16135475
- [Background] Lancee J, van den Bout J, van Straten A, Spoormaker VI. Internet-delivered or mailed self-help treatment for insomnia?: a randomized waiting-list controlled trial. Behav Res Ther. 2012 Jan;50(1):22-9. doi: 10.1016/j.brat.2011.09.012. Epub 2011 Oct 24. PMID 22055281
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Espie CA, Inglis SJ, Harvey L. Predicting clinically significant response to cognitive behavior therapy for chronic insomnia in general medical practice: analysis of outcome data at 12 months posttreatment. J Consult Clin Psychol. 2001 Feb;69(1):58-66. doi: 10.1037//0022-006x.69.1.58. PMID 11302278
- [Background] Espie CA, MacMahon KM, Kelly HL, Broomfield NM, Douglas NJ, Engleman HM, McKinstry B, Morin CM, Walker A, Wilson P. Randomized clinical effectiveness trial of nurse-administered small-group cognitive behavior therapy for persistent insomnia in general practice. Sleep. 2007 May;30(5):574-84. doi: 10.1093/sleep/30.5.574. PMID 17552372
- [Background] Espie CA, Fleming L, Cassidy J, Samuel L, Taylor LM, White CA, Douglas NJ, Engleman HM, Kelly HL, Paul J. Randomized controlled clinical effectiveness trial of cognitive behavior therapy compared with treatment as usual for persistent insomnia in patients with cancer. J Clin Oncol. 2008 Oct 1;26(28):4651-8. doi: 10.1200/JCO.2007.13.9006. Epub 2008 Jun 30. PMID 18591549
- [Background] Kyle SD, Miller CB, Rogers Z, Siriwardena AN, Macmahon KM, Espie CA. Sleep restriction therapy for insomnia is associated with reduced objective total sleep time, increased daytime somnolence, and objectively impaired vigilance: implications for the clinical management of insomnia disorder. Sleep. 2014 Feb 1;37(2):229-37. doi: 10.5665/sleep.3386. PMID 24497651
- [Background] Espie CA, Kyle SD, Hames P, Gardani M, Fleming L, Cape J. The Sleep Condition Indicator: a clinical screening tool to evaluate insomnia disorder. BMJ Open. 2014 Mar 18;4(3):e004183. doi: 10.1136/bmjopen-2013-004183. PMID 24643168
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Derived] Mayo NE, Brouillette MJ, Fellows LK; Positive Brain Health Now Investigators. Understanding and optimizing brain health in HIV now: protocol for a longitudinal cohort study with multiple randomized controlled trials. BMC Neurol. 2016 Jan 14;16:8. doi: 10.1186/s12883-016-0527-1. PMID 26762403